CLINICAL TRIAL: NCT02925598
Title: AuraGainTM and I-Gel® Laryngeal Masks in General Anesthesia for Laparoscopic Cholecystectomy - Performance Characteristics and Effects on Hemodynamics
Brief Title: AuraGainTM and I-Gel® Laryngeal Masks in General Anesthesia for Laparoscopic Cholecystectomy
Acronym: AILMALC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ülkü Sabuncu, Principal Investigator, Ulku Sabuncu, MD, Anesthesiology and Reanimation, Adiyaman University Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2015/178
Record Dates: First submitted 2016-09-05; First posted 2016-10-06 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Aspiration of Gastric Content
Keywords: Laringeal masks; Cholecystectomy, Laparascopic; Intubation, intratracheal

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- I-gel LMA (Experimental): I-gel LMA insertion: I-gel insertion was done in supine position and with a standard gel pillow with the patient's head on following anesthesia induction. The insertion was verified with the manual ventilation of the patient and EtCO2 waveform.
  Interventions: Device: I-gel LMA insertion
- AuraGain LMA (Experimental): AuraGain insertion:AuraGain LMA insertion was done in supine position and with a standard gel pillow with the patient's head on following anesthesia induction. The insertion was verified with the manual ventilation of the patient and EtCO2 waveform.
  Interventions: Device: AuraGain LMA insertion
- Endotracheal tube (ETT) (Experimental): Endotracheal tube insertion: Endotracheal tube (ETT) insertion was done in supine position and with a standard gel pillow with the patient's head on following anesthesia induction. The insertion was verified with the manual ventilation of the patient and EtCO2 waveform.
  Interventions: Device: ETT insertion

INTERVENTIONS:
Device: I-gel LMA insertion — 'I-gel LMA insertion' was done following anesthesia induction.
  Arms: I-gel LMA
Device: AuraGain LMA insertion — 'AuraGain LMA insertion' was done following anesthesia induction.
  Arms: AuraGain LMA
Device: ETT insertion — 'ETT insertion' was done following anesthesia induction.
  Arms: Endotracheal tube (ETT)

SUMMARY:
The standard procedure used for airway control in general anesthesia for LC (laparoscopic cholecystectomy) is endotracheal intubation (EI). AuraGain and I-Gel are supraglottic airway devices (SADs) used for airway control for certain types of surgeries. The aim of this study was to evaluate and compare the performances of new types of SADs with EI regarding their insertion times, durations, perioperative complications and effects on hemodynamic parameters and peak airway pressures (Paw) in LC as well.

DETAILED DESCRIPTION:
The standard procedure used for airway control in general anesthesia for LC (laparoscopic cholecystectomy) is endotracheal intubation (EI). AuraGain and I-Gel are supraglottic airway devices (SADs) used for airway control for certain types of surgeries.Previous studies have investigated and/or compared the performance of ProSeal™ LMA (Intavent Orthofix, Maidenhead, UK) during LC. But the performances of I-Gel and AuraGain have not been studied well yet. The main aim of this study was to evaluate and compare the performances of new types of SADs (i.e. AuraGain and I-Gel) with endotracheal intubation regarding their insertion times, ease of insertion and perioperative complications. The secondary aim was to observe their effects on hemodynamic parameters and peak airway pressures.

ELIGIBILITY:
Inclusion Criteria:

* (ASA) 1-2 physical status scheduled for elective LC

Exclusion Criteria:

* under the age of 18, history of hiatus hernia, gastroesophageal reflux, body mass index (BMI) > 30 kg m-2, ASA physical status 3 or over and patients who met the difficult intubation criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Insertion time | Perioperative
  It was assessed that how many secs it takes to insert the device
Attempts to insertion | Perioperative
  It was assessed that how many attempts needed to insert the device
Airway related complications | Perioperative
  Airway related complications like bronchospasm,gastric regurgitation,smooth tissue damages were assessed

SECONDARY OUTCOMES:
Heart Rate bpm | Perioperative
  Heart rates changes were evaluated preoperative and after device insertion and then in every 5 mins.
Systolic blood pressure mmHg | Perioperative
  Systolic blood pressure changes were evaluate preoperative,following device insertion then in every 5 mins.
Diastolic blood pressure mmHg | Perioperative
  Diastolic blood pressures were evaluated preoperative,following device insertion then in every 5 mins.
Peak airway pressure | Perioperative
  During the surgery peak airway pressures were assessed following device insertion snd then in every 5 mins.

CONTACTS AND LOCATIONS:
Overall Officials: Ulku Sabuncu, MD, Principal Investigator — Adiyaman university Research and Educational Hospital

IPD SHARING:
Plan to Share IPD: No